CLINICAL TRIAL: NCT05586490
Title: Development of a Multifunctional Rehabilitation Standing and Stepping Device for Persons With Parkinson's Disease
Brief Title: Development of a Multifunctional Rehabilitation Device for Persons With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Chatkaew Pongmala, Research Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00216022a; 1R41NS1129418 (Other Grant/Funding Number: NINDS)
Record Dates: First submitted 2022-10-12; First posted 2022-10-19 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease
Keywords: feasibility device testing
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: The feasibility study will involve a sequential stage of device feasibility testing with the initial aims 1 and 2 being a single group and the in-home feasibility testing will involve controls persons for an exploratory data collection. The same participants are asked to proceed sequentially through the three phase of the study. Participants in the third sub-study will then be asked to complete the open label extension.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- In-lab and in home feasibility testing of research device in people with Parkinson's disease (PwP) (Experimental): Multifunctional rehabilitation device for PwP for human user acceptance testing for 2 lab sessions (aim 1) and 5 lab sessions (aim 2). This arm will use the experimental device in home feasibility testing (aim 3). This arm will be asked to participate in the open label extension.
  Interventions: Device: Multifunctional RehabilitationDevice (MRD)
- In-home feasibility testing (alternate device) (Active Comparator): Multifunctional rehabilitation device for PwP for human user acceptance testing for 2 lab sessions (aim 1) and 5 lab sessions (aim 2).
  This arm will use another device to compare to the experimental device for in home feasibility of using the device at home (aim 3). This arm will be asked to participate in the open label extension.
  Interventions: Device: Multifunctional RehabilitationDevice (MRD); Device: existing standard rehabilitation device
- In-home feasibility testing (no device in at home portion) (Other): Multifunctional rehabilitation device for PwP for human user acceptance testing for 2 lab sessions (aim 1) and 5 lab sessions (aim 2). For the at home portion, this arm will not use any device but have the same outcomes measured. (aim 3)
  Interventions: Device: Multifunctional RehabilitationDevice (MRD)

INTERVENTIONS:
Device: Multifunctional RehabilitationDevice (MRD) — Multifunctional rehabilitation device to treat mobility and cognitive problems in PwP
  Other Names: MRD
Device: existing standard rehabilitation device — existing standard rehabilitation device to be used for in-home comparison testing for aim 3
  Arms: In-home feasibility testing (alternate device)

SUMMARY:
The researchers have developed a multifunctional rehabilitation device that will be tested in this feasibility trial across three sub-studies: (i) dual session in-lab; (ii) multi-session in-lab and (iii) in the participant's home. A long-term outcome is to test possible benefits of this device (if accepted by the user Parkinson population) on motor and cognitive functions in a clinical trial in a future study. Participants who receive a device during the in-home trial will have the option to keep the device for up to two years in an open label extension. During this extension, participants can optionally provide feedback on their user experience such as discomfort.

DETAILED DESCRIPTION:
The primary purpose of this feasibility study is to assess human user acceptance of the device during 2 lab sessions (aim 1) from which the persons will proceed to 5 lab sessions (aim 2) and during in-home use (aim 3). The in-home aim will also include control persons to allow exploratory collection of clinical data that may provide preliminary outcome data to properly power a future phase 2 randomized clinical trial. The open label extension will provide information on the efficacy of using the device long-term.

While 45 persons may appear to be a larger than normal number for a device feasibility trial, because Parkinsons patients have a wide range of clinical symptoms, in order to acquire any meaningful data, some "spread" must be achieved. For example, 3 individuals in several different symptomatic categories. Further, there is some chance of attrition. Lastly, to be clear, details of device design may continue to be modified throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease
* Willing and able to comply with study requirements

Exclusion Criteria:

* Parkinson's disease dementia
* Parkinsonism plus syndromes
* Inability to stand, step, or walk without an assistive device
* History of symptoms in stance that preclude safe and comfortable participation, such as severe dizziness and lightheadedness, severe orthostasis, severe symptomatic leg or back musculoskeletal pain, painful neuropathy, significant ankle edema, or medication side effects
* History of symptomatic cardiovascular or pulmonary disease interfering with stance
* History of active rheumatic arthritis
* History of uncontrolled chronic pain syndrome
* Any other history of medical or psychiatric comorbidity precluding safe participation in the project
* Venous stasis or severe varicosities

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chatkaew Pongmala, PhD, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was originally intended to be completed as a sequence from Aim 1 to Aim 2, then to Aim 3. However, due to scheduling conflicts and attrition, subjects were invited to participate in individual aims to ensure sufficient data collection for each aim. Since some subjects completed multiple aims while others completed all aims, results were analyzed by aim, and thus are presented in that way here. In total, 38 participants were enrolled, with 1 withdrawal prior to randomization.
Pre-assignment Details: Of the 37 unique participants who started study procedures, 29 participated in only one aim of the study, while 8 participated in multiple. Of the 8 participants who participated in multiple aims, 2 participants started procedures for aims 1 and 2 only, 3 participants started aims 1 and 3 only, 1 participant started aims 2 and 3 only, and 2 participants started all 3 aims.
Groups:
- Participants Whose 1st Participation Was in Aim 1: Aim 1 consisted of 2-sessions of in-lab feasibility testing of research device in people with Parkinson disease(PwP)
- Participants Whose First Participation Was in Aim 2: Aim 2 consists of 5-sessions of in-lab feasibility testing of research device in people with Parkinson disease(PwP)
  Multifunctional RehabilitationDevice (MRD): Multifunctional rehabilitation device to treat mobility and cognitive problems in PwP
- Participants Whose 1st Participation Was in Aim 3: In-Home Testing - Research Device Arm: Participants of the in-home feasibility trial who were randomized into the research device group. This group includes some participants who also participated in Aims 1 or 2 but dual enrollment did not play a role in analysis of this arm
- Participants Whose 1st Participation Was in Aim 3: In-Home Testing - Alternate Device Arm: Participants of the in-home feasibility trial who were randomized into the alternate device group. This group includes some participants who also participated in Aims 1 or 2 but dual enrollment did not play a role in analysis of this arm
  Multifunctional RehabilitationDevice (MRD): Multifunctional rehabilitation device to treat mobility and cognitive problems in PwP
- Participants Whose 1st Participation Was in Aim 3: In-Home Testing - No Device Arm: Participants of the in-home feasibility trial who were randomized into the no device group. This group includes some participants who also participated in Aims 1 or 2 but dual enrollment did not play a role in analysis of this arm
Period: Completed Data Collection for Aim 1
Arm/Group | Participants Whose 1st Participation Was in Aim 1 | Participants Whose First Participation Was in Aim 2 | Participants Whose 1st Participation Was in Aim 3: In-Home Testing - Research Device Arm | Participants Whose 1st Participation Was in Aim 3: In-Home Testing - Alternate Device Arm | Participants Whose 1st Participation Was in Aim 3: In-Home Testing - No Device Arm
Started | 18 | 0 | 0 | 0 | 0
Completed | 18 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Completed Data Collection for Aim 2
Arm/Group | Participants Whose 1st Participation Was in Aim 1 | Participants Whose First Participation Was in Aim 2 | Participants Whose 1st Participation Was in Aim 3: In-Home Testing - Research Device Arm | Participants Whose 1st Participation Was in Aim 3: In-Home Testing - Alternate Device Arm | Participants Whose 1st Participation Was in Aim 3: In-Home Testing - No Device Arm
Started | 4 | 4 | 0 | 0 | 0
Completed | 4 | 4 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Completed Aim 3 - Research Device Arm
Arm/Group | Participants Whose 1st Participation Was in Aim 1 | Participants Whose First Participation Was in Aim 2 | Participants Whose 1st Participation Was in Aim 3: In-Home Testing - Research Device Arm | Participants Whose 1st Participation Was in Aim 3: In-Home Testing - Alternate Device Arm | Participants Whose 1st Participation Was in Aim 3: In-Home Testing - No Device Arm
Started | 1 | 1 | 5 | 0 | 0
Completed | 1 | 1 | 4 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Period: Completed Aim 3 - Alternate Device Arm
Arm/Group | Participants Whose 1st Participation Was in Aim 1 | Participants Whose First Participation Was in Aim 2 | Participants Whose 1st Participation Was in Aim 3: In-Home Testing - Research Device Arm | Participants Whose 1st Participation Was in Aim 3: In-Home Testing - Alternate Device Arm | Participants Whose 1st Participation Was in Aim 3: In-Home Testing - No Device Arm
Started | 2 | 0 | 0 | 5 | 0
Completed | 1 | 0 | 0 | 5 | 0
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Period: Completed Aim 3 - No Device Arm
Arm/Group | Participants Whose 1st Participation Was in Aim 1 | Participants Whose First Participation Was in Aim 2 | Participants Whose 1st Participation Was in Aim 3: In-Home Testing - Research Device Arm | Participants Whose 1st Participation Was in Aim 3: In-Home Testing - Alternate Device Arm | Participants Whose 1st Participation Was in Aim 3: In-Home Testing - No Device Arm
Started | 2 | 0 | 0 | 0 | 5
Completed | 1 | 0 | 0 | 0 | 5
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants could complete any combination of aims for this study. 37 unique individuals in total participated in the study, 29 of which participated in a single aim, and 8 of which participated in more than one aim. 6 participants participated in 2 aims, and 2 participants participated in all 3 aims. The "Overall Number of Baseline Participants" represents the TOTAL number of participants to participate in each aim while baseline characteristics are reported according to participant FIRST aim.
Groups:
- Participants Whose 1st Participation Was in Aim 1: Multifunctional rehabilitation device for PwP for human user acceptance testing for 2 lab sessions.
- Participants Whose First Participation Was in Aim 2: Multifunctional rehabilitation device for PwP for human user acceptance testing for 5 lab sessions.
- Participants Whose 1st Participation Was in Aim 3: In-Home Testing - Alternate Device Arm: Participants of the in-home feasibility trial who were randomized into the alternate device group. This group includes some participants who also participated in Aims 1 or 2 but dual enrollment did not play a role in analysis of this arm.
- Total: Total of all reporting groups
Arm/Group | Participants Whose 1st Participation Was in Aim 1 | Participants Whose First Participation Was in Aim 2 | Participants Whose 1st Participation Was in Aim 3: In-Home Testing - Research Device Arm | Participants Whose 1st Participation Was in Aim 3: In-Home Testing - Alternate Device Arm | Participants Whose 1st Participation Was in Aim 3: In-Home Testing - No Device Arm | Total
Number analyzed (Participants) | 18 | 8 | 7 | 7 | 7 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Of the 37 unique participants who started study procedures, 29 participated in only one aim of the study, while 8 participated in multiple. Of the 8 participants who participated in multiple aims, 2 participants started procedures for aims 1 and 2 only, 3 participants started aims 1 and 3 only, 1 participant started aims 2 and 3 only, and 2 participants started all 3 aims.
  years
    Completed Data Collection for Aim 1: number analyzed (Participants) | 18 | 0 | 0 | 0 | 0 | 18
    Completed Data Collection for Aim 1 | 71.23 (7.94) |  |  |  |  | 71.23 (7.94)
    Completed Data Collection for Aim 2: number analyzed (Participants) | 4 | 4 | 0 | 0 | 0 | 8
    Completed Data Collection for Aim 2 | 68 (11.8) | 70.75 (6.90) |  |  |  | 69.38 (9.07)
    Completed Data Collection for Aim 3: number analyzed (Participants) | 5 | 1 | 5 | 5 | 5 | 21
    Completed Data Collection for Aim 3 | 71.8 (3.27) | 68 (0) | 65.2 (4.87) | 68.6 (5.68) | 67.6 (5.90) | 68.29 (5.09)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Of the 37 unique participants who started study procedures, 29 participated in only one aim of the study, while 8 participated in multiple. Of the 8 participants who participated in multiple aims, 2 participants started procedures for aims 1 and 2 only, 3 participants started aims 1 and 3 only, 1 participant started aims 2 and 3 only, and 2 participants started all 3 aims.
  Participants
    Completed Data Collection for Aim 1: number analyzed (Participants) | 18 | 0 | 0 | 0 | 0 | 18
    Completed Data Collection for Aim 1: Female | 4 |  |  |  |  | 4
    Completed Data Collection for Aim 1: Male | 14 |  |  |  |  | 14
    Completed Data Collection for Aim 2: number analyzed (Participants) | 4 | 4 | 0 | 0 | 0 | 8
    Completed Data Collection for Aim 2: Female | 0 | 2 |  |  |  | 2
    Completed Data Collection for Aim 2: Male | 4 | 2 |  |  |  | 6
    Completed Data Collection for Aim 3: number analyzed (Participants) | 5 | 1 | 5 | 5 | 5 | 21
    Completed Data Collection for Aim 3: Female | 2 | 1 | 1 | 3 | 2 | 9
    Completed Data Collection for Aim 3: Male | 3 | 0 | 4 | 2 | 3 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Of the 37 unique participants who started study procedures, 29 participated in only one aim of the study, while 8 participated in multiple. Of the 8 participants who participated in multiple aims, 2 participants started procedures for aims 1 and 2 only, 3 participants started aims 1 and 3 only, 1 participant started aims 2 and 3 only, and 2 participants started all 3 aims.
  Participants
    Completed Data Collection for Aim 1: number analyzed (Participants) | 18 | 0 | 0 | 0 | 0 | 18
    Completed Data Collection for Aim 1: Hispanic or Latino | 0 |  |  |  |  | 0
    Completed Data Collection for Aim 1: Not Hispanic or Latino | 18 |  |  |  |  | 18
    Completed Data Collection for Aim 1: Unknown or Not Reported | 0 |  |  |  |  | 0
    Completed Data Collection for Aim 2: number analyzed (Participants) | 4 | 4 | 0 | 0 | 0 | 8
    Completed Data Collection for Aim 2: Hispanic or Latino | 0 | 0 |  |  |  | 0
    Completed Data Collection for Aim 2: Not Hispanic or Latino | 4 | 4 |  |  |  | 8
    Completed Data Collection for Aim 2: Unknown or Not Reported | 0 | 0 |  |  |  | 0
    Completed Data Collection for Aim 3: number analyzed (Participants) | 5 | 1 | 5 | 5 | 5 | 21
    Completed Data Collection for Aim 3: Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
    Completed Data Collection for Aim 3: Not Hispanic or Latino | 5 | 1 | 5 | 5 | 5 | 21
    Completed Data Collection for Aim 3: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Of the 37 unique participants who started study procedures, 29 participated in only one aim of the study, while 8 participated in multiple. Of the 8 participants who participated in multiple aims, 2 participants started procedures for aims 1 and 2 only, 3 participants started aims 1 and 3 only, 1 participant started aims 2 and 3 only, and 2 participants started all 3 aims.
  Participants
    Completed Data Collection for Aim 1: number analyzed (Participants) | 18 | 0 | 0 | 0 | 0 | 18
    Completed Data Collection for Aim 1: American Indian or Alaska Native | 0 |  |  |  |  | 0
    Completed Data Collection for Aim 1: Asian | 0 |  |  |  |  | 0
    Completed Data Collection for Aim 1: Native Hawaiian or Other Pacific Islander | 0 |  |  |  |  | 0
    Completed Data Collection for Aim 1: Black or African American | 0 |  |  |  |  | 0
    Completed Data Collection for Aim 1: White | 18 |  |  |  |  | 18
    Completed Data Collection for Aim 1: More than one race | 0 |  |  |  |  | 0
    Completed Data Collection for Aim 1: Unknown or Not Reported | 0 |  |  |  |  | 0
    Completed Data Collection for Aim 2: number analyzed (Participants) | 4 | 4 | 0 | 0 | 0 | 8
    Completed Data Collection for Aim 2: American Indian or Alaska Native | 0 | 0 |  |  |  | 0
    Completed Data Collection for Aim 2: Asian | 0 | 0 |  |  |  | 0
    Completed Data Collection for Aim 2: Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  |  | 0
    Completed Data Collection for Aim 2: Black or African American | 0 | 0 |  |  |  | 0
    Completed Data Collection for Aim 2: White | 4 | 4 |  |  |  | 8
    Completed Data Collection for Aim 2: More than one race | 0 | 0 |  |  |  | 0
    Completed Data Collection for Aim 2: Unknown or Not Reported | 0 | 0 |  |  |  | 0
    Completed Data Collection for Aim 3: number analyzed (Participants) | 5 | 1 | 5 | 5 | 5 | 21
    Completed Data Collection for Aim 3: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Completed Data Collection for Aim 3: Asian | 0 | 0 | 0 | 0 | 0 | 0
    Completed Data Collection for Aim 3: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Completed Data Collection for Aim 3: Black or African American | 0 | 0 | 0 | 0 | 0 | 0
    Completed Data Collection for Aim 3: White | 5 | 1 | 5 | 5 | 5 | 21
    Completed Data Collection for Aim 3: More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Completed Data Collection for Aim 3: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: Some participants were recruited to participate in more than one aim of the study. "Overall Number of Baseline Participants" represents the total number of individuals enrolled in each arm. The number analyzed here represents the total number of participants whose FIRST participation was in each respective arm.
  Participants
    United States: number analyzed (Participants) | 18 | 4 | 5 | 5 | 5 | 37
    United States | 18 | 4 | 5 | 5 | 5 | 37
(Aim 3) Mean time to complete the Timed Up and Go test (TUG) [Mean (Standard Deviation); unit: seconds] — Mobility test that evaluates the amount of time it takes the participants to stand, walk 3 meters, turn around, walk, and sit back down. Improved performance is indicated by lower time to complete measured in seconds. Population: Only participant data from the Aim 3 arms were analyzed for this measure. In each arm of Aim 3, 1 participant withdrew from the study prior to testing. The Number Analyzed for this measure represents the TOTAL number of participants to undergo this testing for Aim 3, regardless of which aim they first participated in.
  seconds
    number analyzed (Participants) | 0 | 0 | 6 | 6 | 6 | 18
    (all) |  |  | 7.65 (1.68) | 7.49 (1.12) | 8.53 (1.94) | 7.89 (1.58)
(Aim 3) Mean time to complete the Instrumented Stand up and Walk Test (iSAW) [Mean (Standard Deviation); unit: seconds] — Mobility test that evaluates the amount of time it takes the participant to walk 10 feet, make a turn around a cone, and return to the starting position. Improved performance is indicated by lower time to complete measured in seconds. Population: Only participant data from the Aim 3 arms were analyzed for this measure. In each arm of Aim 3, 1 participant withdrew from the study prior to testing. The Number Analyzed for this measure represents the TOTAL number of participants to undergo this testing for Aim 3, regardless of which aim they first participated in.
  seconds
    number analyzed (Participants) | 0 | 0 | 6 | 6 | 6 | 18
    (all) |  |  | 13.05 (1.42) | 12.75 (1.81) | 13.32 (2.02) | 13.03 (1.75)
(Aim 3) Sensory postural control domain as measured during the MiniBESTest. [Mean (Standard Deviation); unit: units on a scale] — Balance test that evaluates how long participants are able to stand on surfaces of varying firmness with eyes open and closed. Domain scores range from 0 to 6 with higher scores indicating stronger sensory postural control. Population: Only participant data from the Aim 3 arms were analyzed for this measure. In each arm of Aim 3, 1 participant withdrew from the study prior to testing. The Number Analyzed for this measure represents the TOTAL number of participants to undergo this testing for Aim 3, regardless of which aim they first participated in.
  units on a scale
    number analyzed (Participants) | 0 | 0 | 6 | 6 | 6 | 18
    (all) |  |  | 5.00 (1.00) | 5.17 (0.37) | 4.33 (1.97) | 4.83 (1.11)
(Aim 3) Mean Movement Disorder Society Unified Parkinson's Disease Rating Scale Part III Score [Mean (Standard Deviation); unit: units on a scale] — The Movement Disorder Society Unified Parkinson's Disease Rating Scale Part 3 (MDS-UPDRS part III) is the motor examination portion of the UPDRS evaluation. Scores range from 0-132, with higher scores indicating greater severity of motor symptoms. Population: Only participant data from the Aim 3 arms were analyzed for this measure. In each arm of Aim 3, 1 participant withdrew from the study prior to testing. The Number Analyzed for this measure represents the TOTAL number of participants to undergo this testing for Aim 3, regardless of which aim they first participated in.
  units on a scale
    number analyzed (Participants) | 0 | 0 | 6 | 6 | 6 | 18
    (all) |  |  | 37.58 (14.61) | 33 (12.06) | 32.25 (10.55) | 34.28 (12.41)
(Aim 3) Mean Modified Hoehn and Yahr stage [Mean (Standard Deviation); unit: units on a scale] — The Hoehn and Yahr scale is a widely used clinical rating scale to categorize the progression of Parkinson's disease into stages ranging no disease (0) to wheelchair bound (5). Population: Only participant data from the Aim 3 arms were analyzed for this measure. In each arm of Aim 3, 1 participant withdrew from the study prior to testing. The Number Analyzed for this measure represents the TOTAL number of participants to undergo this testing for Aim 3, regardless of which aim they first participated in.
  units on a scale
    number analyzed (Participants) | 0 | 0 | 6 | 6 | 6 | 18
    (all) |  |  | 2.17 (0.41) | 1.92 (0.53) | 2.17 (0.61) | 2.09 (0.53)
(Aim 3) Mean response time during the Stroop Stepping Test [Mean (Standard Deviation); unit: seconds] — During this test, subjects make steps based on congruent (stimulus prompts the stepping response) and incongruent (stimulus prompts inhibition of the stepping response) arrows and sounds. These responses are combined to compare the response time for stepping from pre and post intervention visits to determine if reaction time improves (indicated by a decrease in response time). Population: Only participant data from the Aim 3 arms were analyzed for this measure. In each arm of Aim 3, 1 participant withdrew from the study prior to testing. The Number Analyzed for this measure represents the TOTAL number of participants to undergo this testing for Aim 3, regardless of which aim they first participated in.
  seconds
    number analyzed (Participants) | 0 | 0 | 6 | 6 | 6 | 18
    (all) |  |  | 2.10 (0.42) | 1.92 (0.34) | 1.99 (0.15) | 2.00 (0.30)
(Aim 3) Mean time taken to complete Stroop Color Word Interference Test [Mean (Standard Deviation); unit: seconds] — During this test, participants read congruent and incongruent colored names of colors. This will be used to compare the number of incorrect responses and the time it takes to complete the test from pre and post intervention visits to determine if inhibitory control improves (indicated by decrease of incorrect responses and completion time). Population: Only participant data from the Aim 3 arms were analyzed for this measure. In each arm of Aim 3, 1 participant withdrew from the study prior to testing. The Number Analyzed for this measure represents the TOTAL number of participants to undergo this testing for Aim 3, regardless of which aim they first participated in.
  seconds
    number analyzed (Participants) | 0 | 0 | 6 | 6 | 6 | 18
    (all) |  |  | 162.25 (62.74) | 168.82 (77.46) | 167.76 (30.60) | 166.28 (56.93)

OUTCOME MEASURES:

1. Primary Outcome: (Aim 1) Mean of User Acceptance Questionnaire (UAQ) Part 1 Total Scores
Description: Completed at 2nd study visit after a 1-hour session using the device. UAQ part 1 assesses potential difficulties experienced while using the device. UAQ part 1 scores range from 0 to 90, with lower scores indicating fewer difficulties experienced.
Time Frame: After 1-hour session using the device
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- In-lab and in Home Feasibility Testing of Research Device in People With Parkinson's Disease (PwP): Multifunctional RehabilitationDevice (MRD): Multifunctional rehabilitation device to treat mobility and cognitive problems in PwP
  for human user acceptance testing for 2 lab sessions (aim 1)
Arm/Group | In-lab and in Home Feasibility Testing of Research Device in People With Parkinson's Disease (PwP)
Number analyzed (Participants) | 18
score on a scale | 7.28 (6.18)

2. Primary Outcome: (Aim 1) Mean of User Acceptance Questionnaire (UAQ) Part 2 Total Scores
Description: Completed at 2nd study visit after a 1-hour session using the device. UAQ part 2 assesses participant preferences for using the device. UAQ part 2 scores range from 0 to 30, with higher scores indicating greater personal preference for using the device.
Time Frame: After 1-hour session using the device
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-lab and in Home Feasibility Testing of Research Device in People With Parkinson's Disease (PwP)
Number analyzed (Participants) | 18
score on a scale | 23.72 (5.12)

3. Primary Outcome: (Aim 1) Mean System Usability Scale (SUS) Total Scores
Description: Completed at 2nd study visit after a 1-hour session using the device. SUS is a questionnaire consisting of 10 Likert-scale questions to assess usability of the device. Benchmarked scores range from 0 to 100, with higher scores indicating better usability of the device.
Time Frame: After 1-hour session using the device
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-lab and in Home Feasibility Testing of Research Device in People With Parkinson's Disease (PwP)
Number analyzed (Participants) | 18
score on a scale | 83.19 (14.09)

4. Primary Outcome: (Aim 2) Change in Mean Time to Complete the Instrumented Timed Up and Go Test (iTUG)
Description: Mobility test that evaluates the amount of time it takes the participants to stand, walk 10 feet, turn around, walk, and sit back down. Improved performance is indicated by lower time to complete measured in seconds.
Time Frame: After 2-week intervention
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | In-lab and in Home Feasibility Testing of Research Device in People With Parkinson's Disease (PwP)
Number analyzed (Participants) | 8
seconds
  Pre-Intervention | 18.761 (5.651)
  Post-Intervention | 18.124 (4.700)
Statistical Analysis 1: Comparison: In-lab and in Home Feasibility Testing of Research Device in People With Parkinson's Disease (PwP); Test type: Other — A comparison is not being made between two different treatment groups; p = 0.429, t-test, 2 sided — A priori threshold for statistical significance is p < 0.05; Paired samples t-test, df = 7; Mean Difference (Net) = -0.6375

5. Primary Outcome: (Aim 2) Change in Mean Duration of Balance During Romberg Test Condition
Description: Balance test that evaluates how long participants are able to stand on a foam pillow before losing balance. Improved performance is indicated by longer balance duration.
Time Frame: After 2-week intervention
Population: Although in participant flow, the 8 participants are divided by what arm they subsequently participated in, within this outcome measure, there is no logical reason to separate them, as they were all testing the same device used in the same manner.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | In-lab and in Home Feasibility Testing of Research Device in People With Parkinson's Disease (PwP)
Number analyzed (Participants) | 8
seconds
  Pre-Intervention | 26.25 (10.61)
  Post-Intervention | 30 (0)
Statistical Analysis 1: Comparison: In-lab and in Home Feasibility Testing of Research Device in People With Parkinson's Disease (PwP); Test type: Other — A comparison is not being made between two different treatment groups; p = 0.351, t-test, 2 sided — A priori threshold for statistical significance was p < 0.05; Paired samples t-test, df = 7; Mean Difference (Net) = 3.75

6. Primary Outcome: (Aim 2) Change in Mean Response Time During the Stroop Stepping Test
Description: During this test, subjects make steps based on congruent (stimulus prompts the stepping response) and incongruent (stimulus prompts inhibition of the stepping response) arrows and sounds. This will be used to compare the mean response time for stepping from pre and post intervention visits to determine if reaction time improves (indicated by a decrease in response time). Mean times include responses to both congruent and incongruent stimuli.
Time Frame: After 2-week intervention
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | In-lab and in Home Feasibility Testing of Research Device in People With Parkinson's Disease (PwP)
Number analyzed (Participants) | 8
seconds
  Pre-Intervention | 1.887 (0.27)
  Post-Intervention | 1.874 (0.42)
Statistical Analysis 1: Comparison: In-lab and in Home Feasibility Testing of Research Device in People With Parkinson's Disease (PwP); Test type: Other — A comparison is not being made between two different treatment groups; p = 0.937, t-test, 2 sided — A priori threshold for statistical significance was p < 0.05; Paired samples t-test, df = 7; Mean Difference (Net) = -0.013

7. Primary Outcome: (Aim 2) Change in Mean of Time Taken to Complete Stroop Color Word Interference Test
Description: During this test, participants read congruent and incongruent colored names of colors. This will be used to compare the number of incorrect responses and the time it takes to complete the test from pre and post intervention visits to determine if inhibitory control improves (indicated by decrease of incorrect responses and completion time).
Time Frame: After 2-week intervention
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | In-lab and in Home Feasibility Testing of Research Device in People With Parkinson's Disease (PwP)
Number analyzed (Participants) | 8
seconds
  Pre-Intervention | 167.51 (55.96)
  Post-Intervention | 152.71 (54.54)
Statistical Analysis 1: Comparison: In-lab and in Home Feasibility Testing of Research Device in People With Parkinson's Disease (PwP); Test type: Other — A comparison is not being made between two different treatment groups; p = 0.044, t-test, 2 sided — A priori threshold for statistical significance was p < 0.05; Paired samples t-test, df = 7; Mean Difference (Net) = -14.80

8. Primary Outcome: (Aim 3) Difference in Effect of Study Intervention on Mean Time to Complete the Instrumented Timed Up and Go Test (iTUG) in Study Device Group Versus Control Groups.
Description: as for outcome 4
Time Frame: After 14-week intervention
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- In-home Feasibility Testing (Alternate Device): Multifunctional rehabilitation device for PwP for human user acceptance testing for 2 lab sessions (aim 1) and 5 lab sessions (aim 2).
  This arm will use another device to compare to the experimental device for in home feasibility of using the device at home (aim 3). This arm will be asked to participate in the open label extension.
  Multifunctional RehabilitationDevice (MRD): Multifunctional rehabilitation device to treat mobility and cognitive problems in PwP
  existing standard rehabilitation device: existing standard rehabilitation device to be used for in-home comparison testing for aim 3
Arm/Group | In-lab and in Home Feasibility Testing of Research Device in People With Parkinson's Disease (PwP) | In-home Feasibility Testing (Alternate Device) | In-home Feasibility Testing (no Device in at Home Portion)
Number analyzed (Participants) | 6 | 6 | 6
seconds
  Pre-Intervention | 7.65 (1.68) | 7.49 (1.12) | 8.53 (1.94)
  Post-Intervention | 8.27 (1.77) | 6.83 (1.42) | 8.47 (2.34)
Statistical Analysis 1: Comparison: In-home Feasibility Testing (Alternate Device) vs In-home Feasibility Testing (no Device in at Home Portion); Test type: Superiority; p = 0.42, ANCOVA — A priori threshold for statistical significance was p < 0.05; Estimated difference between groups (alternate device and no device group) controlling for pre-trial measurements, gender, and age; Mean Difference (Net) = -0.68
Statistical Analysis 2: Comparison: In-lab and in Home Feasibility Testing of Research Device in People With Parkinson's Disease (PwP) vs In-home Feasibility Testing (no Device in at Home Portion); Test type: Superiority; p = 0.50, ANCOVA — A priori threshold for statistical significance was p < 0.05; Estimated difference between groups (research device group and no device group) controlling for pre-trial measurements, gender, and age; Mean Difference (Net) = 0.57

9. Primary Outcome: (Aim 3) Difference in Effect of Intervention on Mean Time to Complete the Instrumented Stand and Walk Test (iSAW) in Study Device Group Versus Control Groups.
Description: Mobility test that evaluates the amount of time it takes the participant to walk 10 feet, make a turn around a cone, and return to the starting position. Improved performance is indicated by lower time to complete measured in seconds.
Time Frame: After 14-week intervention
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | In-lab and in Home Feasibility Testing of Research Device in People With Parkinson's Disease (PwP) | In-home Feasibility Testing (Alternate Device) | In-home Feasibility Testing (no Device in at Home Portion)
Number analyzed (Participants) | 6 | 6 | 6
seconds
  Pre-Intervention | 13.05 (1.42) | 12.72 (1.81) | 13.32 (2.02)
  Post-Intervention | 12.40 (1.76) | 11.35 (1.99) | 11.92 (2.21)
Statistical Analysis 1: Comparison: In-home Feasibility Testing (Alternate Device) vs In-home Feasibility Testing (no Device in at Home Portion); Test type: Superiority; p = 0.986, ANCOVA — A priori threshold for statistical significance was p < 0.05; [statistical method as in outcome 8, analysis 1]; Mean Difference (Net) = -0.03
Statistical Analysis 2: Comparison: In-lab and in Home Feasibility Testing of Research Device in People With Parkinson's Disease (PwP) vs In-home Feasibility Testing (no Device in at Home Portion); Test type: Superiority; p = 0.479, ANCOVA — A priori threshold for statistical significance was p < 0.05; Estimated difference between groups (research device and no device group) controlling for pre-trial measurements, gender, and age; Mean Difference (Net) = -1.25

10. Primary Outcome: (Aim 3) Difference in Effect of Intervention on Sensory Postural Control Domain as Measured During the MiniBESTest.
Description: Balance test that evaluates how long participants are able to stand on surfaces of varying firmness with eyes open and closed. Domain scores range from 0 to 6 with higher scores indicating stronger sensory postural control.
Time Frame: After 14-week intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-lab and in Home Feasibility Testing of Research Device in People With Parkinson's Disease (PwP) | In-home Feasibility Testing (Alternate Device) | In-home Feasibility Testing (no Device in at Home Portion)
Number analyzed (Participants) | 6 | 6 | 6
units on a scale
  Pre-Intervention | 5.00 (1.00) | 5.17 (0.37) | 4.33 (1.97)
  Post-Intervention | 3.83 (1.46) | 4.5 (1.71) | 3.33 (1.60)
Statistical Analysis 1: Comparison: In-home Feasibility Testing (Alternate Device) vs In-home Feasibility Testing (no Device in at Home Portion); Test type: Superiority; p = 0.098, ANCOVA — A priori threshold for statistical significance was p < 0.05; [statistical method as in outcome 8, analysis 1]; Mean Difference (Net) = -0.195
Statistical Analysis 2: Comparison: In-lab and in Home Feasibility Testing of Research Device in People With Parkinson's Disease (PwP) vs In-home Feasibility Testing (no Device in at Home Portion); Test type: Superiority; p = 0.729, ANCOVA — A priori threshold for statistical significance was p < 0.05; [statistical method as in outcome 9, analysis 2]; Mean Difference (Net) = -0.039

11. Primary Outcome: (Aim 3) Difference in Effect of Intervention on Mean Movement Disorder Society Unified Parkinson's Disease Rating Scale Part III Score in Study Device Group Versus Control Groups.
Description: Movement Disorder Society Unified Parkinson's Disease Rating Scale Part 3 (MDS-UPDRS part III) is the motor examination portion of the UPDRS evaluation. Scores range from 0-132, with higher scores indicating greater severity of motor symptoms.
Time Frame: After 14-week intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-lab and in Home Feasibility Testing of Research Device in People With Parkinson's Disease (PwP) | In-home Feasibility Testing (Alternate Device) | In-home Feasibility Testing (no Device in at Home Portion)
Number analyzed (Participants) | 6 | 6 | 6
score on a scale
  Pre-Intervention | 37.58 (14.61) | 33 (12.06) | 32.25 (10.55)
  Post-Intervention | 36.83 (12.91) | 27.67 (8.86) | 36.58 (9.55)
Statistical Analysis 1: Comparison: In-home Feasibility Testing (Alternate Device) vs In-home Feasibility Testing (no Device in at Home Portion); Test type: Superiority; p = 0.0580, ANCOVA — A priori threshold for statistical significance was p < 0.05; [statistical method as in outcome 8, analysis 1]; Mean Difference (Net) = -8.15
Statistical Analysis 2: Comparison: In-lab and in Home Feasibility Testing of Research Device in People With Parkinson's Disease (PwP) vs In-home Feasibility Testing (no Device in at Home Portion); Test type: Superiority; p = 0.718, ANCOVA — A priori threshold for statistical significance was p < 0.05; [statistical method as in outcome 9, analysis 2]; Mean Difference (Net) = -1.54

12. Primary Outcome: (Aim 3) Mean Modified Hoehn and Yahr Stage at Baseline
Description: The Hoehn and Yahr scale is a widely used clinical rating scale to categorize the progression of Parkinson's disease into stages ranging no disease (0) to wheelchair bound (5).
Time Frame: At baseline (descriptive statistic)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-lab and in Home Feasibility Testing of Research Device in People With Parkinson's Disease (PwP) | In-home Feasibility Testing (Alternate Device) | In-home Feasibility Testing (no Device in at Home Portion)
Number analyzed (Participants) | 6 | 6 | 6
score on a scale | 2.17 (0.41) | 1.92 (0.58) | 2.17 (0.61)

13. Primary Outcome: (Aim 3) Difference in Effect of Intervention on Response Time During the Stroop Stepping Test in Study Device Group Versus Control Groups.
Description: During this test, subjects make steps based on congruent (stimulus prompts the stepping response) and incongruent (stimulus prompts inhibition of the stepping response) arrows and sounds. These responses are combined to compare the response time for stepping from pre and post intervention visits to determine if reaction time improves (indicated by a decrease in response time). Mean times include responses to both congruent and incongruent stimuli.
Time Frame: After 14-week intervention
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | In-lab and in Home Feasibility Testing of Research Device in People With Parkinson's Disease (PwP) | In-home Feasibility Testing (Alternate Device) | In-home Feasibility Testing (no Device in at Home Portion)
Number analyzed (Participants) | 6 | 6 | 6
seconds
  Pre-Intervention | 2.10 (0.42) | 1.92 (0.34) | 1.99 (0.15)
  Post-Intervention | 1.92 (0.50) | 1.83 (0.33) | 1.97 (0.33)
Statistical Analysis 1: Comparison: In-home Feasibility Testing (Alternate Device) vs In-home Feasibility Testing (no Device in at Home Portion); Test type: Superiority; p = 0.816, ANCOVA — A priori threshold for statistical significance was p < 0.05; [statistical method as in outcome 8, analysis 1]; Mean Difference (Net) = 0.063
Statistical Analysis 2: Comparison: In-lab and in Home Feasibility Testing of Research Device in People With Parkinson's Disease (PwP) vs In-home Feasibility Testing (no Device in at Home Portion); Test type: Superiority; p = 0.985, ANCOVA — A priori threshold for statistical significance was p < 0.05; [statistical method as in outcome 9, analysis 2]; Mean Difference (Net) = -0.0048

14. Primary Outcome: (Aim 3) Difference in Effect of Study Device Intervention on Time Taken to Complete Stroop Color Word Interference Test in Study Device Group Versus Control Groups.
Description: as for outcome 7
Time Frame: After 14-week intervention
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | In-lab and in Home Feasibility Testing of Research Device in People With Parkinson's Disease (PwP) | In-home Feasibility Testing (Alternate Device) | In-home Feasibility Testing (no Device in at Home Portion)
Number analyzed (Participants) | 6 | 6 | 6
seconds
  Pre-Intervention | 162.25 (62.74) | 168.82 (77.46) | 167.76 (30.60)
  Post-Intervention | 158.53 (63.42) | 163.19 (72.97) | 153.95 (20.57)
Statistical Analysis 1: Comparison: In-home Feasibility Testing (Alternate Device) vs In-home Feasibility Testing (no Device in at Home Portion); Test type: Superiority; p = 0.59, ANCOVA — A priori threshold for statistical significance was p < 0.05; [statistical method as in outcome 8, analysis 1]; Mean Difference (Net) = 6.33
Statistical Analysis 2: Comparison: In-lab and in Home Feasibility Testing of Research Device in People With Parkinson's Disease (PwP) vs In-home Feasibility Testing (no Device in at Home Portion); Test type: Superiority; p = 0.51, ANCOVA — A priori threshold for statistical significance was p < 0.05; [statistical method as in outcome 9, analysis 2]; Mean Difference (Net) = 8.16

ADVERSE EVENTS:
Time Frame: For the randomized portion, data was collected for the 12 weeks of device testing. But for those participants who were involved in lab testing , data would be gathered over 1 week (2 visits) for those involved in substudy 1, and over 2 weeks for those involved in substudy 2.
Description: Adverse event data are presented according to each aim of the study. There was 1 arm for both aims 1 and 2, and 3 arms for aim 3. Some subjects participated in multiple aims.
Groups:
- Aim 1: 2-session In-lab Feasibility Testing of Research Device in People With Parkinson Disease(PwP): Multifunctional rehabilitation device for PwP for human user acceptance testing for 2 lab sessions.
- Aim 2: 5-session In-lab Feasibility Testing of Research Device in People With Parkinson Disease(PwP): Multifunctional rehabilitation device for PwP for human user acceptance testing for 5 lab sessions.
- Aim 3: In-home Feasibility Testing - Research Device Arm: Participants of the in-home feasibility trial who were randomized into the research device group. This group includes some participants who also participated in Aims 1 or 2 but dual enrollment did not play a role in analysis of this arm.
- Aim 3: In-home Feasibility Testing - Alternate Device Arm: Participants of the in-home feasibility trial who were randomized into the alternate device group. This group includes some participants who also participated in Aims 1 or 2 but dual enrollment did not play a role in analysis of this arm
- Aim 3: In-home Feasibility Testing - No Device Arm: Participants of the in-home feasibility trial who were randomized into the no device group. This group includes some participants who also participated in Aims 1 or 2 but dual enrollment did not play a role in analysis of this arm.
Arm/Group | Aim 1: 2-session In-lab Feasibility Testing of Research Device in People With Parkinson Disease(PwP) | Aim 2: 5-session In-lab Feasibility Testing of Research Device in People With Parkinson Disease(PwP) | Aim 3: In-home Feasibility Testing - Research Device Arm | Aim 3: In-home Feasibility Testing - Alternate Device Arm | Aim 3: In-home Feasibility Testing - No Device Arm
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/8 | 0/7 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/8 | 0/7 | 0/7 | 1/7
Other Adverse Events (participants affected / at risk) | 1/18 | 0/8 | 7/7 | 6/7 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aim 1: 2-session In-lab Feasibility Testing of Research Device in People With Parkinson Disease(PwP) (N=18) | Aim 2: 5-session In-lab Feasibility Testing of Research Device in People With Parkinson Disease(PwP) (N=8) | Aim 3: In-home Feasibility Testing - Research Device Arm (N=7) | Aim 3: In-home Feasibility Testing - Alternate Device Arm (N=7) | Aim 3: In-home Feasibility Testing - No Device Arm (N=7)
Transient ischemic attack (TIA) (Vascular disorders) | 0 | 0 | 0 | 0 | 1 (1) — Unrelated to study, serious and unexpected AE.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aim 1: 2-session In-lab Feasibility Testing of Research Device in People With Parkinson Disease(PwP) (N=18) | Aim 2: 5-session In-lab Feasibility Testing of Research Device in People With Parkinson Disease(PwP) (N=8) | Aim 3: In-home Feasibility Testing - Research Device Arm (N=7) | Aim 3: In-home Feasibility Testing - Alternate Device Arm (N=7) | Aim 3: In-home Feasibility Testing - No Device Arm (N=7)
Fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 — Probably related, mild, expected AE
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 2 | 2 — Probably related, mild, expected AE
Dizziness (Cardiac disorders) | 0 | 0 | 2 | 1 | 0 — Related, mild, expected AE
Intercurrent Illness (General disorders) | 0 | 0 | 1 | 2 (3) | 1 — Unrelated, mild, unexpected AE
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 — Related, mild, expected AE
Eye Strain (Eye disorders) | 0 | 0 | 0 | 1 | 0 — Unrelated, mild, unexpected AE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT05586490/Prot_SAP_001.pdf
  • Informed Consent Form (2023-08-17): https://cdn.clinicaltrials.gov/large-docs/90/NCT05586490/ICF_000.pdf